CLINICAL TRIAL: NCT06002087
Title: Unified Protocol for Transdiagnostic Treatment: An Adaptation and Pilot RCT for the Treatment of Depression and Anxiety in Adults
Brief Title: Unified Protocol for Transdiagnostic Treatment for Depression and Anxiety in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Science and Technology, Pakistan (Other)
Responsible Party: Principal Investigator, Asma Nisa, Primary Researcher, National University of Science and Technology, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0988/Ethic/01/S3H/083/DBS
Record Dates: First submitted 2023-08-03; First posted 2023-08-21 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Depression; Anxiety
Keywords: Anxiety; Depression; Emotion Regulation; Evidence-Based Treatment; Transdiagnostic
MeSH Terms: conditions — Depression; Anxiety Disorders; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Experimental group: Participants in the experimental group will receive the Unified Protocol (UP) treatment.
  Control group: Participants in the control group will be placed on a waitlist and will not receive any treatment until the end of the study.
Masking Description: To ensure blinding of participants and intervention facilitator, a randomizing researcher, who is different from the facilitator, will generate the sequences and assign an ID (1-50) to one of the groups based on the sequence. The sealed envelopes will be given to the facilitator, who will open the envelope in the interview and inform the participants about their allocated group. This will ensure that neither the participants nor the facilitator will know which group they are assigned to, which will help to minimize bias in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group: Unified Protocol (UP) (Experimental): Participants will receive 14 weekly individual sessions of 50-60 minutes each using the adapted UP treatment.
  Interventions: Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders
- Control group: Waitlist Control (No Intervention): Participants in the control group will be placed on a waitlist and will not receive any treatment until the end of the study.

INTERVENTIONS:
Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders — The current researchers adapted the Unified Protocol (UP) treatment and used the adapted version in this study. UP outlines two complimentary modules for goal setting and psychoeducation followed by five core treatment modules: mindful emotion awareness, cognitive flexibility, countering emotional behaviors, awareness and tolerance of physical sensations, and emotion exposures, and an optional relapse prevention module to help people maintain their gains after treatment.
  Other Names: UP
  Arms: Experimental group: Unified Protocol (UP)

SUMMARY:
To conduct a pilot randomized controlled trial (RCT) of a culturally adapted Unified Protocol (UP) for transdiagnostic psychological treatment in adults (age 18 and above) with anxiety and/or depression to assess the feasibility and acceptability of UP treatment.

The main questions it aims to answer are:

1. To assess the estimates of likely recruitment rates including how many approached, volunteered, screened, retained, and complete the treatment and what is the dropout rate?
2. To what degree do participants adhere and engage with the treatment procedures?
3. To what extent do the participants feel satisfied with the treatment?
4. To what degree do participants complete self-report and clinician-administered measures of anxiety, depression, functional impairment, and emotion regulation?
5. What is the treatment outcome with regard to emotion regulation, symptoms of anxiety, depression, functional impairment, and emotion regulation?

The participants will be randomized to either the treatment group or the control group. The treatment group will receive 14 sessions of one-on-one individual treatment with the Unified Protocol. The control group will receive no treatment.

DETAILED DESCRIPTION:
Most patients with depression and anxiety in low-resource settings don't get evidence-based treatment. Transdiagnostic approaches like UP are promising for these settings because they are multi-problem, modular, flexible, and have low complexity. The present study aimed to investigate the initial acceptability and feasibility of the adapted Unified Protocol (UP) in relation to its quantitative and qualitative effects on attendance, homework compliance, satisfaction, and perceived usefulness of the intervention. Additionally, the study aimed to evaluate the preliminary effects of the adapted UP on depression, anxiety, functional impairment, and emotion regulation among adults suffering from anxiety, depression, and/or comorbidity of both disorders.

A sample size of approximately 50 adults will be recruited from mental health facilities and online dissemination of the study. After screening through the Beck Depression Inventory-II (BDI-II) and Beck Anxiety Inventory (BAI), and assessing the inclusion and exclusion criteria, those who demonstrate moderate to severe scores on the BDI-II and BAI will be further evaluated by the principal investigator using the Structured Clinical Interviews for DSM-5 (Research Version) (SCID-5-RV) to determine their diagnosis. Once the eligibility criteria are met, participants will be randomly assigned to one of two study conditions:

Experimental group: Participants in the experimental group will receive the Unified Protocol (UP) treatment.

Control group: Participants in the control group will be placed on a waitlist and will not receive any treatment until the end of the study.

Participants from both groups will complete several assessment measures at baseline, mid-treatment (only at week 7 of the UP), and post-treatment.

To ensure protocol quality and fidelity, the therapist has a master's degree in Clinical Psychology and two years of previous supervised clinical experience in cognitive behavioral therapy (CBT). The therapist also participated in introductory and intermediate-level training workshops for the Unified Protocol (UP) and received UP Therapist Certification. The therapist has received supervision from the UP-certified psychologist and received 18 weeks of individualized supervision on a course of treatment utilizing the UP. Weekly supervision sessions were conducted via video-conferencing (Zoom), and transcripts of the sessions were reviewed for adherence to the protocol and competence in protocol delivery throughout the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* suffering from anxious and/or depressive disorder

Exclusion Criteria:

* suicide risk at the time of assessment
* comorbidity of pervasive developmental disorder
* comorbidity of psychotic disorders
* severe physical illness
* receiving concurrent psychotherapy
* receiving psychopharmacological treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Feasibility- Recruitment method | 14 weeks
  The number of participants recruited by each of the three methods used for recruiting. The methods will be: mental health facilities, online dissemination, and referrals and recommendations.
Feasibility- Recruitment rate | 14 weeks
  To assess the estimates of likely recruitment rates, including:
  How many participants approached? How many participants volunteered? How many participants were screened? How many participants were retained in the study? What was the dropout rate? The number of participants completing the final assessment (assessed through a record made at each session).
Feasibility- Weekly face-to-face sessions | 14 weeks
  The nature of barriers that may lead to participants dropping out of treatment can be assessed by examining the number and type of problems that they experienced while attending weekly sessions. These problems include transportation difficulties, work or educational demands, childcare difficulties, scheduling conflicts, and treatment procedures interfering with daily life. Followed by an open-ended question that will assess any other reason to discontinue the treatment.
Feasibility: Eligibility criteria | 14 weeks
  Assessed through the number of participants fulfilling the eligibility criteria from the total number of participants registered, number of ineligible participants, and reasons for ineligibility.
Feasibility - Treatment adherence and engagement | 14 weeks
  Engagement in treatment will be assessed using the Homework Rating Scale-Revised, a 12-item measure that assesses beliefs, consequences, and engagement with treatment homework activities. Total scores range from 0 to 48 on this scale, where higher scores indicate higher commitment to the treatment. Treatment adherence will be further assessed by tracking participant attendance, percentage of intervention completion, and number of sessions completed.
Feasibility - Semi-structured Interview for treatment adherence and engagement | 14 weeks
  Semi-structured questions will be asked by an independent interviewer to assess the reasons for adherence and non-adherence to the treatment.
Acceptability of randomization | 14 weeks
  The number of participants who consented to randomization, number of participants who refused, and reasons for refusal.
Acceptability of the treatment | 14 weeks
  It will be measured through client satisfaction questionnaire. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Acceptability of the treatment - Semi-structured interview | 14 weeks
  Semi-structured interview by an independent interviewer will be conducted to obtain responses on a number of indicators including; Participants' overall satisfaction with the treatment, understand the overall content covered in the treatment, the perceived usefulness of the techniques learned, the discomfort it generated, the likelihood that participants would choose such a treatment again, their recommendation to friends or family, what they found most, what they find least helpful, any modifications they would recommend.
Feasibility of outcome measures | 14 weeks
  Feasibility of outcome measures will be assessed through the assessment completion rates by participants.

SECONDARY OUTCOMES:
Beck Depression Inventory-II | 14 weeks
  It is a 21-item self-report questionnaire to assess depressive symptoms with scores ranging from 0 to 3. Higher scores indicate worse depressive symptoms.
Beck Anxiety Inventory | 14 weeks
  It is a 21-item self-report questionnaire to assess the severity of anxiety symptoms with scores ranging from 0 to 3. Higher scores indicate worse anxiety symptoms.
Work and Social Adjustment Scale | 14 weeks
  It represents a simple measurement of impairment of functioning and consists of 5 items, each rated on an 8-point severity scale adding up to a maximum severity of 40 points. It is validated for use across the full spectrum of psychiatric disorders.
Difficulties in Emotion Regulation Scale | 14 weeks
  It is a 36-item scale with 6 subscales that measure emotion dysregulation and emotional self-regulation strategies. The subscales are non-acceptance of emotional responses, difficulty in performing purposeful behavior, difficulty controlling impulse, lack of emotional awareness, limited access to emotion regulation strategies, and lack of clarity of emotion. The items are scored on a scale of 1 to 5, with higher scores indicating more severe difficulties in emotion regulation.
Positive and Negative Affect Schedule | 14 weeks
  It is a self-report measure that assesses the two broad dimensions of affect: positive affect and negative affect. It is a 20-item scale, and items are rated on a 5-point scale, with higher scores indicating higher experience of those emotions.

OTHER OUTCOMES:
Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders-5, the Research Version | 14 weeks
  The Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders-5 is a semi-structured interview guide for making the major Diagnostic and Statistical Manual of Mental Disorders-5 diagnoses. The current study is using this scale to ensure that all of the study subjects have symptoms that meet the DSM-5 criteria for Major Depressive Disorder and/or anxiety disorder and that all of the subjects with Substance Use Disorder, Bipolar Disorder, or Psychotic Disorders are excluded. The items are scored on a scale of 1 to 3. A higher score on this scale suggests the presence of a mental condition.

CONTACTS AND LOCATIONS:
Overall Officials: Salma Siddiqui, Study Chair — National University of Science and Technology, Pakistan; Amantia A. Ametaj, Study Director — Harvard School of Public Health (HSPH)
Locations (1):
- National University of Sciences and Technology, Pakistan, Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No